CLINICAL TRIAL: NCT03957746
Title: Set Volume of Optimal Resistance Exercise to Generate Hypotension in Hypertensive Elderly Subjects: a Crossover Study
Brief Title: Set Volume of Optimal Resistance Exercise to Generate Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, José Casaña Granell, Director, PhD, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 000018819
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Hypertension; Post-Exercise Hypotension; Resistance Training
MeSH Terms: conditions — Hypertension; Post-Exercise Hypotension | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3 sets of resistance exercise (Experimental)
  Interventions: Other: Resistance training
- 6 sets of resistance exercise (Experimental)
  Interventions: Other: Resistance training
- 9 sets of resistance exercise (Experimental)
  Interventions: Other: Resistance training
- Rest (No Intervention)

INTERVENTIONS:
Other: Resistance training — 3, 6 or 9 sets of biceps curl with elastic bands at 20 repetition-maximum (RM)
  Arms: 3 sets of resistance exercise; 6 sets of resistance exercise; 9 sets of resistance exercise

SUMMARY:
This study evaluates the volume of optimal resistance exercise to generate postexercise hypotension after performing a single exercise in hypertensive elderly subjects. 20 subjects will perform 1 control session and 3 resistance training sessions with different volume: 3, 6 and 9 sets

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive subjects treated with antihypertensive medication
* Controlled blood pressure
* Age between 55 and 70 years old
* Sedentary (less than 150 minutes per week of moderate physical activity and/or 75 minutes per week of vigorous physical activity)
* Non-smokers
* Non-alcoholics
* Informed consent

Exclusion Criteria:

* Any kidney, lung, neurological or psychiatric disease
* Unable to perform exercises
* Participation in other physical activity programs during the study or in the previous 3 months

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Baseline
Blood pressure | Immediately after the end of resistance training session
Blood pressure | 30 minutes after the end of resistance training session
Blood pressure | 60 minutes after the end of resistance training session
Blood pressure | 4 hours after the end of resistance training session
Blood pressure | 5 hours after the end of resistance training session
Blood pressure | 6 hours after the end of resistance training session

SECONDARY OUTCOMES:
Heart rate | Baseline
Heart rate | Immediately after the end of resistance training session
Heart rate | 30 minutes after the end of resistance training session
Heart rate | 60 minutes after the end of resistance training session
Heart rate | 4 hours after the end of resistance training session
Heart rate | 5 hours after the end of resistance training session
Heart rate | 6 hours after the end of resistance training session

CONTACTS AND LOCATIONS:
Overall Officials: Jose Casaña, Principal Investigator — University of Valencia; Joaquín Calatayud, Study Chair — University of Valencia; Alba Cuerda, Study Chair — University of Valencia
Locations (1):
- Primary Health-Care Center, Rocafort, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gargallo P, Casana J, Suso-Marti L, Cuenca-Martinez F, Lopez-Bueno R, Andersen LL, Lopez-Bueno L, Cuerda-Del Pino A, Calatayud J. Minimal Dose of Resistance Exercise Required to Induce Immediate Hypotension Effect in Older Adults with Hypertension: Randomized Cross-Over Controlled Trial. Int J Environ Res Public Health. 2022 Oct 31;19(21):14218. doi: 10.3390/ijerph192114218. PMID 36361100